CLINICAL TRIAL: NCT03465007
Title: Effects of Corticosteroids on Intra-dialytic Hypotension
Brief Title: Steroids on Intra-dialytic Hypotension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Jordan (Other)
Responsible Party: Principal Investigator, Saif Aldeen AlRyalat, Researcher, University of Jordan
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: JUH2018_3
Record Dates: First submitted 2018-03-06; First posted 2018-03-14 (Actual); Last update posted 2019-04-08 (Actual); Status verified 2019-04

CONDITIONS: Dialysis Hypotension
Keywords: hemodialysis; cortisol; Hydrocortisone
MeSH Terms: interventions — Hydrocortisone; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Hydrocortisone (Active Comparator): 100mg Hydrocortisone will be administered prior to hemodialysis
  Interventions: Drug: Hydrocortisone
- Placebo (Placebo Comparator): 100mg normal saline will be administered prior to hemodialysis
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Hydrocortisone — we will give IV Hydrocortisone 100 mg prior to HD to the patients who developed intra-dialytic hypotension and monitor their BP response during the HD treatments.
  Arms: Hydrocortisone
Drug: Normal saline — we will give IV normal saline 100 mg prior to HD to the patients who developed intra-dialytic hypotension and monitor their BP response during the HD
  Arms: Placebo

SUMMARY:
Symptomatic hypotension during (or immediately following) hemodialysis complicates 5 to 30 percent of all dialysis treatments and is associated with increased morbidity and mortality. Kidney Disease Outcomes Quality Initiative (KDOQI) and European Best Practice Guidelines define intradialytic hypotension as the presence of a decrease in systolic blood pressure ≥20 mmHg or a decrease in mean arterial pressure by 10 mmHg, providing the decrease in blood pressure is associated with clinical events and need for nursing interventions. Common causes of intradialytic hypotension include excessive or rapid ultrafiltration, high blood flow during dialysis, CHF, taking the antihypertensive medications prior to HD, and others. One of the possible reasons that is surprisingly has not been approached worldwide for intra-dialytic hypotension could be more prevalent adrenal insufficiency in ESRD patients or a delay in the appropriate rise of endogenous serum cortisol given hemodialysis is considered by all means a stressful condition to the body. Investigators will assess first the prevalence of intradialytic hypotension at JUH dialysis unit. Investigators will screen patients who developed intradialytic hypotension for adrenal insufficiency by ordering random am cortisol. Then Investigators will give IV Hydrocortisone 100 mg prior to HD to patients who developed intra-dialytic hypotension and monitor their BP response during the HD treatments for 3 HD sessions (1 week, 3 HD sessions). After that, the same patients will receive 100 mg normal saline for 3 HD sessions. Both the administrator and the patient will be blinded for the interventions.

ELIGIBILITY:
Inclusion Criteria:

* Patients on hemodialysis who develop intra-dialytic hypotension.

Exclusion Criteria:

* Adrenal insufficiency

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2017-10-22 (Actual); Primary Completion 2018-07-25 (Actual); Study Completion 2019-02-01 (Actual)

PRIMARY OUTCOMES:
Intra-dialytic hypotension | 3 months
  intradialytic hypotension as the presence of a decrease in systolic blood pressure ≥20 mmHg or a decrease in mean arterial pressure by 10 mmHg.

CONTACTS AND LOCATIONS:
Locations (1):
- School of Medicine, Amman, Jordan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Alhawari HH, Alshelleh S, Alhawari HH, Alawwa IA, AlRyalat SA, Mesmar A, Ojjoh K, Alzoubi KH. Effect of Hydrocortisone on Intradialytic Hypotension: A Preliminary Investigational Study. Biomed Res Int. 2020 May 5;2020:4987547. doi: 10.1155/2020/4987547. eCollection 2020. PMID 34901264